CLINICAL TRIAL: NCT06069531
Title: Effect of Oral Probiotic Heat-killed Lactobacillus Johnsonii TCI250 or White Pomegranate Extract on the Vaginal Flora
Brief Title: Effect of Lactobacillus Johnsonii or White Pomegranate Extract on the Vaginal Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: TCI Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shih Chien Huang, assistant professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS1-22188
Record Dates: First submitted 2023-10-02; First posted 2023-10-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Vaginitis Bacterial; Inflammation, Ear
Keywords: Bacterial Vaginitis; Probiotics; white pomegranate extract; Inflammation; Vaginal flora
MeSH Terms: conditions — Vaginosis, Bacterial; Otitis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus johnsonii, (Placebo Comparator): heat-killed Lactobacillus johnsonii TCI250
  Interventions: Dietary Supplement: Lactobacillus johnsonii, Placebo Comparator: White pomegranate extract
- White pomegranate extract (Experimental): White pomegranate extract, dosage of 500mg
  Interventions: Dietary Supplement: Lactobacillus johnsonii, Placebo Comparator: White pomegranate extract

INTERVENTIONS:
Dietary Supplement: Lactobacillus johnsonii, Placebo Comparator: White pomegranate extract — Group A: Placebo; Group B: heat-killed Lactobacillus johnsonii TCI250; Group C: White pomegranate extract, dosage of 500mg for 8 weeks.
  Other Names: Group A: Placebo; Group B: heat-killed Lactobacillus johnsonii TCI250; Group C: White pomegranate extract

SUMMARY:
The goal of this clinical trial is to explore the effect of Lactobacillus johnsonii and white pomegranate extract on female bacterial status, it aims to answer are:

* Evaluate Lactobacillus johnsonii TCI250 probiotics or white pomegranate extract in regulating female vaginal bacteria and improving vaginal health.
* Evaluate Lactobacillus johnsonii TCI250 probiotics or white pomegranate extract in regulating inflammation.

Participants will be randomly assigned to placebo (n = 50), probiotic heat-killed Lactobacillus johnsonii TCI250 group (n = 50) and white pomegranate extract group (n = 50) for 8 weeks. Researchers will compare the vaginal flora and inflammation.

DETAILED DESCRIPTION:
This study is an interventional trial conducted in a randomized double-blind controlled study, we will recruit 150 participants. Participants will be randomly d divided into three groups (Group A: Placebo; Group B: heat-killed Lactobacillus johnsonii TCI250; Group C: White pomegranate extract, dosage of 500mg) for 8 weeks. Subsequently, participants will be followed up for an additional 8 weeks to observe changes in the vaginal microbiota and inflammation. At weeks 0, 4, 8, and 16, participants will record basic information such as personal dietary habits, lifestyle, and health conditions. Additionally, vaginal epithelial cells and whole blood (5 mL) will be collected at weeks 0, 8, and 16 for liver and kidney function monitoring (GPT, creatinine).

1. Study Participants i. Inclusion Criteria (1) Females aged 20-45 (2) Nugent score ≥ 4 (3) Menstrual cycle of 28-60 days ii. Exclusion Criteria (1) Pregnant or lactating women (2) Antibiotic usage (3) Other reproductive-related inflammatory diseases (e.g., candidiasis, gonorrhea, chlamydia infection) (4) Allergy to probiotics or White Pomegranate-related components

   iii. Withdrawal Criteria Participants are free to decide whether to participate in this trial, and they can withdraw their consent at any time during the trial without providing any reason. If participants experience discomfort, they may withdraw from the trial at any time without facing any penalties or compromising their rights.
2. Subject Recruitment Interested participants will be recruited openly through posters posted at Chung Shan Medical University Hospital. The researchers will explain the trial content for 15-20 minutes, and if interested, participants will sign the informed consent form.
3. Research Methods i. Questionnaire assessment ii. Nugent score evaluation iii. Inflammatory markers detection: Including IL-4, IL-10, IL-6, IL-8, MCP-1, TNF-α, IL-1β. I iv. Microbiota gene sequencing: Utilizing 16S rRNA gene sequences to analyze the vaginal microbiota.
4. Statistical Methods Data from this study will be analyzed using SigmaPlot statistical software (version 12.5; Systat Software, San Jose, CA) and SAS statistical software (version 9.4, Statistical Analysis System Institute Inc., Cary, NC, USA). One-way ANOVA will be used to compare differences among the three groups, repeated measurement ANOVA to compare pre- and post-intervention values within each group, and multiple linear regression to analyze the impact of supplement intake on vaginitis scores, inflammation, and microbiota diversity. The results will be presented as mean ± standard deviation (SD). Statistical significance will be indicated by p < 0.05.

Through this study, the administration of Lactobacillus johnsonii TCI250 probiotics and White Pomegranate extract is investigated for their effectiveness in improving the vaginal microbiota in women. This could potentially serve as a means of promoting vaginal health and well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 20-45
2. Nugent score ≥ 4
3. Menstrual cycle of 28-60 days

Exclusion Criteria:

1. Pregnant or lactating women
2. Antibiotic usage
3. Other reproductive-related inflammatory diseases (e.g., candidiasis, gonorrhea, chlamydia infection)
4. Allergy to probiotics or White Pomegranate-related components

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiota | 16 weeks
  Utilizing 16S rRNA gene sequences to analyze the vaginal microbiota, Expecting to increase the proportion of lactobacilli and decrease the proportion of Gardnerella in vaginal.

SECONDARY OUTCOMES:
Nugent score | 16 weeks
  The Nugent Score (0-10) is a Gram-stain scoring system for vaginal swabs for diagnosing bacterial vaginosis (BV). A score of 0 to 3 are considered negative for BV, 4-6 are considered BV-intermediate, and 7-10 are considered to indicate BV. This study anticipates a significant reduction in scores after supplementation, which signifies an improvement in BV.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No